CLINICAL TRIAL: NCT03210831
Title: Clinical Model for Early Predictors of Necrotizing Enterocolitis in Neonates
Brief Title: Early Predictors of Necrotizing Enterocolitis in Neonates
Status: Recruiting | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Oluyinka Olutoye, MD, PhD, Principal Investigator, Nationwide Children's Hospital
Other Study IDs: NCH-00000631
Record Dates: First submitted 2017-07-05; First posted 2017-07-07 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-05

CONDITIONS: Necrotizing Enterocolitis
Keywords: NEC, tissue oxygenation, gut inflammation
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, urine and stools samples are collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this project is to identify neonates who are predisposed to Necrotizing Enterocolitis (NEC). the investigators will determine the effectiveness of non-invasive measures as well as biochemical markers to identify neonates early in the disease process. Thus, the investigators aim to identify infants with NEC prior to the onset of symptoms to institute or test treatments in the long term to prevent the progression of the disease in these infants.

DETAILED DESCRIPTION:
The study will enroll premature, low birth weight infants in the Neonatal Intensive Care Units (NICU). Potential study subjects will be identified upon delivery, or transfer to the NICU, and notification by the neonatology service. Infants born at less than 30 weeks gestational age, birth weight less than or equal to 1500 grams will be eligible for enrollment in the study. The purpose of the study designed is to compare the splanchnic tissue oxygenation index and gut inflammatory biomarkers of patients with any stage of NEC with healthy controls. Since we will not be able to determine which patients will develop NEC a priori, we will anticipate enrolling up to 450 neonates to identify 15 neonates with NEC.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at ≤30 weeks gestational age and/or
* Infants with a birth weight ≤1500 grams

Exclusion Criteria:

* gestational age at birth greater than 30 weeks
* obvious dysmorphic syndromes
* any abdominal wall defect including omphalocele or gastroschisis
* any known intestinal atresia
* complex cardiac abnormalities
* any known lethal chromosomal abnormalities

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: low birth weight, preterm infants
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2017-09-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
splanchnic tissue oxygenation in population at high risk for NEC | 2026
  splanchnic tissue oxygenation as a predictor of NEC

CONTACTS AND LOCATIONS:
Overall Officials: Oluyinka Olutoye, MD, PhD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided